CLINICAL TRIAL: NCT06930300
Title: Vasopressin in the Elderly: Physiological Changes in Neuroendocrine Function and Urinary Secretion in Healthy Aging
Acronym: VENUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2025-00474
Record Dates: First submitted 2025-03-25; First posted 2025-04-16 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Healthy Ageing
MeSH Terms: interventions — Sodium Chloride; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation first, Suppression second (Experimental)
  Interventions: Other: Hypertonic 3% saline; Other: Water
- Suppression first, Stimulation second (Experimental)
  Interventions: Other: Hypertonic 3% saline; Other: Water

INTERVENTIONS:
Other: Hypertonic 3% saline — Participants receive 10 ml/kg body weight of 3% saline infused over 1 hour. The aim is to stimulate copeptin release.
Other: Water — Participants ingest 20 ml/kg water over 1h. The aim is to suppress copeptin release.

SUMMARY:
Elderly people are at a high risk for disturbances in water homeostasis, with both hypo- and hypernatremia being more common with increasing age. Several changes in the physiology of the ageing body are responsible for this predisposition towards hypo- and hypernatremia, including diminished thirst perception, decreasing kidney function, and altered body composition. In addition, age-related changes in AVP secretion have been suggested, but findings remain inconclusive. Possibly, this controversy is due to measurement challenges of AVP.

Copeptin, a surrogate marker of AVP-release, is more stable and a reliable assay is commercially available. While copeptin stimulation and suppression has been studied in healthy volunteers, no study assessed possible changes in copeptin dynamics occurring with ageing.

Therefore, the aim of this study is to investigate copeptin levels in hypo- and hyperosmolar states in generally healthy elderly adults compared to young controls. The investigators hypothesize that both the suppression and stimulation of copeptin is impaired and that the overall range of variation is diminished with increasing age.

This is a monocentric open-labeled randomized controlled trial conducted at the university hospital Basel. All participants will be scheduled for a copeptin stimulation test using hypertonic saline infusion and a copeptin suppression test using water ingestion. The order of the two study visits will be randomized at study inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years or ≥ 60 years
* Normonatremia (135-145 mmol/L)
* Plasma osmolality 280-300 mOsm/kg
* BMI ≥18 and ≤ 30 kg/m2

Exclusion Criteria:

* Regular use of medication with effects on water homeostasis (e.g. blood pressure medication, neuroleptics, desmopressin, etc.)
* Any severe disease requiring frequent medical care, except physiotherapy and/or psychotherapy
* Pacemaker or ICD
* History of thrombosis
* Active oncologic disease
* Heart failure
* Liver cirrhosis
* Estimated glomerular filtration rate (eGFR) < 60 ml/kg/1.73 m2
* Uncontrolled hypertension >160 mmHg systolic or >100 mmHg diastolic
* Polydipsia (ingestion of >3L fluids per day) and polyuria (>50 ml/kg urine production within 24 hours)
* Pregnancy or breastfeeding
* Participation in a study with investigational drugs within 30 days
* Acute illness
* Inability to follow study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — male female
Enrollment: 32 (Actual)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Range of Variation in Copeptin | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, and 120 minutes both after saline administration and after water ingestion
  The primary outcome is the range of variation in copeptin, i.e. difference of suppressed copeptin to the stimulated copeptin, in healthy elderly participants compared to young controls.

SECONDARY OUTCOMES:
Changes in Copeptin upon stimulation and suppression | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Differences in total body water (L) measured by body impedance analysis | at Baseline
Changes in cortisol (mmol/L) | Baseline, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in blood pressure (mmHg) | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in heart rate | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in plasma sodium (mmol/L) | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in plasma potassium (mmol/L) | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in plasma chloride (mmol/L) | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in plasma osmolality (mOsm/kg) | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in estimated glomerular filtration rate (ml/kg/1.73m2) | Baseline, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in plasma glucose (mmol/L) | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in plasma urea (mmol/L) | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in plasma uric acid (umol/L) | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in urine osmolality (mOsm/kg) | Baseline, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in urine sodium (mmol/L) | Baseline, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in urine potassium (mmol/L) | Baseline, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in urine chloride (mmol/L) | Baseline, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in urine urea (mmol/L) | Baseline, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in urine uric acid (umol/L) | Baseline, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in urine glucose (mmol/L) | Baseline, 60 minutes, and 120 minutes both after saline administration and after water ingestion
Changes in urine creatinine (umol/L) | Baseline, 60 minutes, and 120 minutes both after saline administration and after water ingestion

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided